CLINICAL TRIAL: NCT04530708
Title: Multicentre Phase III Study: Addition of Radiotherapy to Standard Medical Treatment for Stage IV NSCLC
Brief Title: Addition of Radiotherapy to Standard Medical Treatment for Stage IV NSCLC
Acronym: MARS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Swedish Lung Cancer Study Group (Network)
Responsible Party: Principal Investigator, Ass. Prof. Jan Nyman, Head of Swedish Lung Cancer Study Group, Ass. Prof., Swedish Lung Cancer Study Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MARS
Record Dates: First submitted 2020-03-27; First posted 2020-08-28 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Radiotherapy; Non Small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer; Quality of Life
Keywords: NSCLC; Radiotherapy; Quality of life
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: Multicentre randomized phase 3 trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A: Standard of care (No Intervention): Normal standard of care and follow-up.
- B: Thoracic radiotherapy (Experimental): Addition of thoracic radiotherapy to 36 Gy after medical treatment.
  Interventions: Radiation: Thoracic radiotherapy

INTERVENTIONS:
Radiation: Thoracic radiotherapy — 36 Gy to the primary lung tumor and present mediastinal node metastases after three months of medical treatment.
  Arms: B: Thoracic radiotherapy

SUMMARY:
The hypothesis for this study is that addition of a moderate dose of radiotherapy to the primary tumor and mediastinal nodes after three months of medical treatment could reduce the tumor burden, partly as an abscopal effect, and thereby improving quality of life and possible also prolonging survival for stage IV NSCLC.

DETAILED DESCRIPTION:
Primary objective: To assess whether the addition of radiotherapy to the remaining thoracic tumor burden following standard medical treatment results in a superior quality of life measured with lung cancer symptom scale (LCSS) in patients with stage IV non-small cell lung cancer. The comparison will be made at three months after randomization.

Secondary objectives: Overall survival, progression-free survival, toxicity and longitudinal quality of life measurements.

Design: Multicentre, randomized, phase III trial. Patients will be registered for the study up-front but randomization will be performed after evaluation of response, three months after initiating medical treatment with chemotherapy/ chemo-immunotherapy or immunotherapy. Randomization will be to thoracic radiotherapy or follow-up (1:1).

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological confirmed non-small cell lung cancer (NSCLC)
* Stage IV disease
* Previously untreated disease (before first line treatment)
* No symptomatic brain metastases
* Performance status (WHO) 0-2
* FEV1 (forced expiratory volume one second) ≥ 1 L or >40% of predicted
* Written informed consent
* Life expectancy ≥ 12 weeks
* Platelet count ≥ 100,00/mm3
* Hemoglobin ≥ 10 g/dl
* WBC (White blod cells) ≥ 3,000/mm3
* Kidney function allowing chemotherapy
* Patients scheduled for standard platinum based chemotherapy, chemo-immunotherapy or immunotherapy
* Willing and able to comply with study treatment

Exclusion Criteria:

* Requirement for daily supplemental oxygen
* Second primary malignancy within 3 years, except for any of the following which can be included even if diagnosed within the past 3 years: Carcinoma in situ of the cervix, nonmelanoma skin cancer, history of low-grade (Gleason score ≤ 6) localized prostate cancer, definitely treated stage I breast cancer, other malignancy that was diagnosed and definitely treated ≥ 3 years ago with no subsequent evidence of recurrence
* Concurrent severe and/or uncontrolled medical condition, including any of the following:
* Angina pectoris
* Congestive heart failure within the past 3 months, unless LVEF (left ventricular ejection fraction) > 40%
* Myocardial infarction within the past 6 months
* Clinically significant infection
* Psychiatric illness or social situation that would limit compliance with study requirements
* EGFR (epidermal growth factor receptor) mutation or ALK (anaplastic lymphoma kinas) - rearrangement detected

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Difference in quality of life | Three months after randomization
  LCSS, lung cancer symptom scale. A scale from zero to one-hundred, higher number indicate worse symptoms.

SECONDARY OUTCOMES:
Overall survival | 24 months
  From randomization
Progression free survival | 24 months
  From randomization
Toxicity of esophagitis, pneumonitis, dyspnea, fatigue, cough | During follow-up , up to 24 months.
  CTC (common toxicity criteria) version 4.0. Esophagitis, pneumonitis, dyspnea, fatigue, cough, worst grade.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Nyman, Ass.prof, Principal Investigator — Sahlgrenska University Hospital; Thomas Björk-Eriksson, Prof., Study Director — Regionalt Cancercentrum Väst
Locations (3):
- Sweden (3):
  - Department of Oncology, Norrlands Universitetssjukhus, Umeå, Norrland
  - Department of Oncology, Karolinska University Hospital, Stockholm, Stockholm County
  - Department of Oncology, Sahlgrenska University Hospital, Gothenburg, Västra Götaland County

DOCUMENTS (1):
  • Study Protocol (2019-10-17): https://cdn.clinicaltrials.gov/large-docs/08/NCT04530708/Prot_000.pdf